CLINICAL TRIAL: NCT05122325
Title: Vibration and Transcutaneous Tibial Nerve Stimulation As a Treatment for Sexual Dysfunction in Women with Spinal Cord Injury: a Randomized Clinical Trial
Brief Title: Treatment for Sexual Dysfunction in Women with Spinal Cord Injury
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Cristina Lirio (Other)
Responsible Party: Sponsor-Investigator, Cristina Lirio, Director, University of Castilla-La Mancha
Organization: University of Castilla-La Mancha (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLirio06
Record Dates: First submitted 2021-11-02; First posted 2021-11-16 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2024-12

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal cord injuries; Women; Pelvic floor disorders; Sexuality
MeSH Terms: conditions — Spinal Cord Injuries; Pelvic Floor Disorders; Sexuality

STUDY DESIGN:
Intervention Model Description: Participants will randomize to three groups: an intervention group 1 contracted transcutaneous electrostimulation through the tibial nerve (n = 18), an intervention group 2 that occurred with genital vibration (n = "18) and a control group (n = 18)
Who Masked: Outcomes Assessor
Masking Description: Blind and concealed randomisation will be performed in assessment and data analysis. The assignment to groups will only be known by the main researcher who will be in charge of indicating in a sealed envelope to care providers and each participant the group to which participants have been assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intervention group 1: Transcutaneous tibial nerve stimulation (TTNS) (Experimental): Transcutaneous application of low frequency electrical current over the tibial nerve TENS® EMS NMS60 for a 30 minutes session, twice a week.
  Placing a small electrode 3 fingers up to the internal malleolus and 1 cm posterior (adjusting its placement with a point finder or testing with low frequencies of 2-3 Hz). A large electrode placed in the calcaneus.
  Interventions: Device: Transcutaneous tibial nerve stimulation TENS® EMS NMS60 device
- Intervention group 2: Genital vibration (Experimental): Women will be instructed in the use of the Ferticare 2.0® vibrator with a frequency of 70 Hz, amplitude of 1.5 mm. It will be recommended to gradually increase its use over time, with a limit of 30 minutes a day.
  Interventions: Device: Genital vibration with Ferticare 2.0® vibrator
- Control group (Sham Comparator): A sham of TTNS intervention with the device turned off, twice a week.
  Interventions: Device: TENS® EMS NMS60 device_sham intervention

INTERVENTIONS:
Device: Transcutaneous tibial nerve stimulation TENS® EMS NMS60 device — Stimulation sessions with a TENS® EMS NMS60 device. These will be carried out for 30 minutes, once a week at 10 Hz, with a pulse width of 200 μs and an intensity between 0 and 100 mA, which will be individually adjusted to each participant.
  Inicially, frequency between 2-3 Hz, so that when the current passes, a contraction-relaxation will cause the first toe movement visually evident (excitomotor threshold).
  Once verified, the frequency is raised to what has been established between 10Hz and there the intensity is increased without having to now reach the excitomotor threshold, as long as the physiotherapist notice it is enough (it must be tolerable).
  Other Names: TTNS
  Arms: Intervention group 1: Transcutaneous tibial nerve stimulation (TTNS)
Device: Genital vibration with Ferticare 2.0® vibrator — Women will be instructed in the use of the Ferticare 2.0® vibrator. Initially, a practice will be carried out , indicating that the frequency of use will be 70 Hz with an amplitude of 1.5 mm. It will be recommended to gradually increase its use over time, with a limit of 30 minutes a day.
  Other Names: vibration
  Arms: Intervention group 2: Genital vibration
Device: TENS® EMS NMS60 device_sham intervention — Sham of TTNS intervention with Stimulation sessions with a TENS® EMS NMS60 device. These will be carried out for 30 minutes, once a week.
  Inicially, frequency between 2-3 Hz, so that when the current passes, a contraction-relaxation will cause the first toe movement visually evident (excitomotor threshold).
  Once verified, the intensity is decreased to lower the sensitive threshold of treatment.
  Other Names: Control
  Arms: Control group

SUMMARY:
Women with spinal cord injury frequently experience sexual dysfunction such as disturbances during arousal and an increased time to orgasm. However, little evidence has been found on its therapeutic approach and low adherence. To verify the effectiveness of two interventions: the application of genital vibration and transcutaneous stimulation of the tibial nerve.

This is a randomized clinical trial. 54 women will be recruited who suffer from sexual dysfunction.

DETAILED DESCRIPTION:
The allocation will be randomly assign to the three groups: an intervention group 1 transcutaneous electrostimulation of tibial nerve (n = 18), an intervention group 2 genital vibration (n = "18) and a control group (n = 18). The treatment time will be 12 weeks. Treatment adherence, as well as treatment effectiveness, will be evaluated through the Female Sexual Function Index, the "Sexual Quality of Life-Female" questionnaire, quantitative sensory tests and the improvement reported by the patient in arousal and orgasm. Evaluations will be carried out before treatment, at the end of the treatment, and at 3 and 6 months after the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Women with incomplete spinal cord injury B, C or D (with preservation of the sacral arch and sensitive assessment of the lower dermatomes not absent, paying special attention to the sensitivity of the genital area) level below T6.
* between 18-60 years
* hormonal analysis. Participants do not present menopausal values of the hormone FSH (follicle stimulating hormone ) (31- 134 U / L)
* present some type of sexual disorder secondary to spinal cord injury with at least 12 months of evolution
* from Spain
* willing to attend the evaluation and treatment center
* seeking to improve in the sexual area.

Exclusion Criteria:

* women with active pregnancy
* present pre-existing pathologies in the genital area
* genital malformation, previous neurosurgery that affects the genital response capacity
* sexual disorders before the injury
* pressure ulcers, serious medical illness or any type of pathology in which the use of sick leave is contraindicated frequency
* psychiatric disorder, narcotic dependence, use of specific serotonin reuptake inhibitors, antipsychotics or other drugs that affect sexual response.
* does not sign the informed consent.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
The "Index of female sexual function (IFSF)" | 5 minutes
  This questionnaire showed validity, internal consistency in all its domains, specifically Cronbach's Alpha 0.745 in arousal and 0.753 in orgasm and test-retest reliability of ICC 0.96. This questionnaire consists of 19 questions and is grouped into six domains. The score for each domain is multiplied by a factor and the final result is the arithmetic sum of the domains. The higher the score, the better sexuality.
Sexual Quality of Life-Female (SQOL-F) | 5 minutes
  SQOL-F showed good validity and reliability. The questionnaire was developed to measure the impact of sexual disorders on quality of life. This questionnaire consists of 18 questions with a response scale of 6 options. The quality of sexual life will be considered poor if the score is between 18-51, moderate between 51-84 and good if it is greater than 84.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Lirio-Romero, PhD, Study Director — University of Castilla-La Mancha
Locations (1):
- Cristina Lirio-Romero, Toledo, Toledo, Spain

IPD SHARING:
Plan to Share IPD: No